CLINICAL TRIAL: NCT01273675
Title: An Investigation on the Effect of Candesartan on Early Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chu-Su, Yu, National Taiwan University Hospital
Other Study IDs: 201008056R
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-09

CONDITIONS: Diabetic Nephropathy
Keywords: Hypertension; Primary disease
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is well understood that hypertension, dyslipidemia, and diabetes mellitus are the major risks of chronic kidney disease. Current guidelines recommend screening kidney estimated glomerular filtration function with serum creatinine. But it is not the utmost effective method and the GFR would be underestimated. Since good correlation was noticed between serum creatinine and chronic kidney disease, urinary microalbumin levels is better for patients with risks of chronic kidney diseases. With adequate and early education, or antihypertensive agents with angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB), all could alleviate renal function deterioration and the severity of proteinuria. As a result, high sensitive methods is urgent and needed for early screening and diseases following up under medication with ACEi and ARB in chronic kidney disease patients. In this project, the investigators are going to include the patients with typy II diabetes mellitus combining with hypertension who are treated with antihypertensive agents. Such volunteers will be treated with Candesartan 8-16mg/ day and maintain systolic blood pressure <130 mm/Hg, diastolic blood pressure < 80 mm/ Hg as the goal. Therefore, this project would make effort on correlation with urinary microalbumin and other biomarkers changes under Candesartan treatment- one of ARB medication for 12 weeks, and further exploration of new biomarkers that may be related to renal parenchymal injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Type II Diabetic disease with hypertension (BP: systolic 140-160 mm/Hg, diastolic 80-100 mm/Hg) for 8 weeks.
2. HbA1c< 8.0%
3. Cre. <1.5 g/dL and eGFR: 89 - 30 mL/min/1.73 m2

Exclusion Criteria:

1. Pregnancy
2. During the observation, BP: systolic >160 mm/Hg, diastolic >100 mm/Hg).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II Diabetic diasese with hypertension ( systolic 140-160 mm/Hg, dystolic 80-100 mm/Hg) for 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chu-Su, PhD candidate, Principal Investigator — National Taiwan University Hospital